CLINICAL TRIAL: NCT06058273
Title: Improvement of the Phonatory Outcome in Patients Undergoing Open Partial Horizontal Laryngectomy (OPHL) and Speech Therapy by Applying the Bruni® Training: a Prospective Cohort Study
Brief Title: Bruni® Training in OPHL Patients
Acronym: BTLS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, LONGOBARDI YLENIA, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5631
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Substitution Voice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OPHL patients (Experimental)
  Interventions: Behavioral: Bruni® training

INTERVENTIONS:
Behavioral: Bruni® training — 10 sessions (7 individual and 3 group) based on the Bruni method, which was born as a method for the artistic voice (rock, pop, gospel, R&B, grunge, metal), acting and dubbing. It is a method based on the didactic desire to lead any artist to the ability to produce various types of noise, specifically generically supraglottic, predominantly arytenoid and falsechordal emissions, providing the perceptive, proprioceptive and praxis tools to safely emit and manage the many sounds generated from a supraglottic source

SUMMARY:
Surgically treated patients with type II OPHL being treated at the Phoniatrics Unit of the Fondazione Policlinico Universitario A. Gemelli-IRCCS, but not satisfied with their voice after the first cycle of therapy with a standard rehabilitation approach, will be recruited. To interested patients, a specific vocal rehabilitation program based on Bruni training will be proposed in order to compare the results obtained using this method with those following the previous treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18;
* Italian mother tongue;
* ability to produce the replacement voice;
* ability to provide written informed consent

Exclusion Criteria:

* < 1 year from the end of both surgical and radiotherapy treatment;
* presence of disease recurrence;
* sensory, neurological deficits
* Learning disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximum phonation time | 3 months
  emit a sustained /a/ for as long as possible with a single air intake. The test will be repeated three times and the longest of the three attempts will be calculated as MPT
type of spectrogram | 3 months
  A sustained /a/ will be recorded, subsequently analyzed with the PRAAT software.
foundamental frequency | 3 months
  A sustained /a/ will be recorded, subsequently analyzed with the PRAAT software
Formantic peaks | 3 months
  The dysillabic word /papà/ will be recorded, subsequently analyzed with the PRAAT software
perceptual evaluation | 3 months
  Voices will be perceptually rated by expert clinicians using the INFVo scale which includes overall impression (I), amount of unintentional additive noise (N), fluency (F) and voice quality (Vo). For each parameter the score can vary from 0 to 10. The higher the score, the better the perceived voice quality.
self evaluation of voice | 3 months
  Patients will be administered the self-evaluation questionnaire "Self-evaluation of Communicative Experience after Laryngeal cancer" which measures adaptation to the replacement voice through 35 items in three subscales (General, Environment, Attitude). Patients should rate each statement on a 4-point categorical scale. You can get a total score from 0 to 102 and three subscores. A score ≥60 suggests the need for specific psychological intervention for acceptance of the new voice.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli - IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No